CLINICAL TRIAL: NCT05285995
Title: The Effect of Two Distraction Strategies in Reducing Preoperative Anxiety in Children：A Randomized Controlled Trial
Brief Title: The Effect of Two Distraction Strategies in Reducing Preoperative Anxiety in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Jie Zhang, Principal investigator, Central South University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: XWANG
Record Dates: First submitted 2022-02-28; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Attention-Distributing Strategies; Preoperative Anxiety
Keywords: Attention-Distributing Strategies; Preoperative Anxiety; Child; Operation

STUDY DESIGN:
Intervention Model Description: In the music group, on the basis of the routine preoperative care, the preferred music was selected from the music library as the intervention content on the day of surgery according to the preference of the children in the 1-day preoperative visit. If there was no preference, the music was played randomly. The children in animation group also chose their favorite cartoons as the intervention content on the basis of preoperative care. During the intervention period, the children in intervention group were also accompanied by a nurse, who was also responsible for the implementation and maintenance of the intervention program.
  The control group received routine care, which included routine preoperative visits and psychological comfort to the children.
Who Masked: Participant, Outcomes Assessor
Masking Description: All patients were screened by researchers for eligibility and then enrolled in the study if eligible and if they provided consent. We divided the subjects into three groups, animation group, music group and control group. According to the 1:1:1 balance of three groups, the statistician set the block length to 3, and carried out a random design of the single-blind block group. According to the sequence of the children entering the study, each group of 3 persons was randomly divided into 3 subjects in each block according to the random number table. The blind copy shall be kept by the personnel of the unit who have nothing to do with the experiment. The randomization plan will be saved by the statistician, and the researcher only has the number of each subject. After opening the envelope according to the number, they know whether the subject is the control group or the intervention group. Investigators involved in the intervention were not involved in the analysis of the study data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The music group (Experimental): In the music group, on the basis of the routine preoperative care, the preferred music was selected from the music library as the intervention content on the day of surgery according to the preference of the children in the 1-day preoperative visit. If there was no preference, the music was played randomly. During the intervention, the same multimedia audio system (Wanderer EDIFIER R1700BT) was used to play music for 30-40 minutes, the volume was controlled at 35-80dB, and adjusted in time according to the feedback of the children.
  Interventions: Other: Music Intervention
- The animation group (Experimental): The children in animation group also chose their favorite cartoons as the intervention content on the basis of preoperative care. The same pad (Lenovo TB3-850F) was used to play pre-selected cartoons, and volume as the music group. During the intervention period, the children in intervention group were also accompanied by a nurse, who was also responsible for the implementation and maintenance of the intervention program.
  Interventions: Other: The animation intervention
- The control group (No Intervention): No interventions except routine preoperative visits and conventional care were performed for the control group.

INTERVENTIONS:
Other: Music Intervention — Before the operation, subjects were asked to choose their favorite music to listen so as to reduce the anxiety before the operation and before the induction of anesthesia.
  Arms: The music group
Other: The animation intervention — Before surgery, subjects were asked to choose their favorite cartoons to watch to reduce anxiety before surgery and induction of anesthesia.
  Arms: The animation group

SUMMARY:
As a very threatening stressor, surgery often leads to strong psychological stress reactions in surgical patients before surgery, the most typical of which is anxiety. According to previous studies, more than 60% of children have severe anxiety during induction of anesthesia. Preoperative anxiety in children is not only significantly related to postoperative adverse physiological and psychological changes such as delirium during recovery from anesthesia, postoperative pain, and sleep disturbance, but also has a serious negative impact on their future study and life (such as timidity, nocturia, etc.), even for several years. Moreover, if the child is uncooperative, crying violently, and refuses to enter the operating room due to preoperative psychological stress, coercive measures are often adopted in clinical practice, which can easily cause harm to the physical and mental health of the child. Therefore, effective interventions to reduce pre-operative anxiety in children is an urgent need.

At present, most researches adopt different interventions to improve the preoperative anxiety of children. Several studies have explored to the efficacy of psychological interventions and virtual reality exposure in reducing preoperative anxiety in children undergoing surgery,results suggest that these interventions can reduce preoperative anxiety and postoperative pain in children. Through toys and video games, researchers verified the effects of psychological preparation on perioperative stress, anxiety, and mood in children undergoing cardiac surgery. In addition, researchers also conducted specialized games, interest induction, childlike and diversified nursing methods to relieve preoperative anxiety in children. Although these interventions have achieved certain effects, the intervention strategies need professionals accompanied and special arrangements, there also exist problems such as time-consuming, labor-intensive, and limited audience, especially during the peak operation period.

Attention distraction is an emotion regulation strategy commonly used in daily life, which actively separates the individual's attention from negative emotions and points to neutral or positive stimuli. Music and animation are the most common and affordable distraction strategies to reduce preoperative anxiety in children, but their effects are inconsistent. It is worth noting that Chow believe that the effect of the combination of audio and video is better than that of music intervention. Moreover, previous studies confirmed that when a mental image is experienced, there is an associated emotion that connects the feeling state with the mind and body leading to a physiologic change.

Therefore, this study intends to use two distraction strategies (music and animation) in pediatric surgery patients to compare the effects of the two strategies on preoperative anxiety, anesthesia induction cooperation, vital signs, and to explore effective methods to improve preoperative anxiety in children.

This study was a randomized controlled trial according to the CONSORT guidelines.Researchers recruited child patients(3-12 years) from a general tertiary hospital in Changsha, Hunan province, China. Researchers divided the subjects into three groups, animation group, music group and control group. The 181 patients recruited were randomized into three groups. Instruments, including preoperative anxiety,the degree of cooperation of children during anesthesia induction ,heart rate and blood pressure were assessed at the three moments: before entering the operating room (baseline T0), entering the operating room(T1), and before induction of anesthesia(T2). The repeated-measures analysis of variance were used to analyze the data.

DETAILED DESCRIPTION:
The study was a single blind, randomized, controlled trial.Researchers recruited subjects from one Central South University-affiliated general tertiary hospital in Changsha, Hunan province, China. And the whole trail was on the basis of the CONSORT statements.Study procedures were approved by the institutional review boards of all participating centers before data collection began. All patients were screened by researchers for eligibility and then enrolled in the study if eligible and if the provided consent.

According to the statistics of the operation center, the main types of operations performed on children are adenoidectomy, tonsillectomy and pediatric occult penile surgery. The literature shows that the age of children undergoing tonsillectomy and adenoidectomy is concentrated in 4-12 years old, and the children with hidden penis surgery are concentrated in 3-12 years old. Therefore, the age for the patients were from 3 to 12 years.Researchers explained the study purposes,procedures, benefits, and risks involved orally to children's parents and participants were recruited with their parents' informed consent.

According to the sequence of the children entering the study, each group(animation group, music group and control group) of 3 persons was randomly divided into 3 subjects in each block according to the random number table. The blind copy shall be kept by the personnel of the unit who have nothing to do with the experiment. The randomization plan will be saved by the statistician, and the researcher only has the number of each subject. After opening the envelope according to the number, the researcher knew whether the subject is the control group or the intervention group. Investigators involved in the intervention were not involved in the analysis of the study data.

In the music group, on the basis of the routine preoperative care, the preferred music was selected from the music library as the intervention content on the day of surgery according to the preference of the children in the 1-day preoperative visit. If there was no preference, the music was played randomly. During the intervention, the same multimedia audio system (Wanderer EDIFIER R1700BT) was used to play music for 30-40 minutes, the volume was controlled at 35-80dB, and adjusted in time according to the feedback of the children.The children in animation group also chose their favorite cartoons as the intervention content on the basis of preoperative care. The same pad (Lenovo TB3-850F) was used to play pre-selected cartoons, and volume as the music group. During the intervention period, the children in intervention group were also accompanied by a nurse, who was also responsible for the implementation and maintenance of the intervention program.

In the control group, the children were received the routine care. One day before the operation, nurses from operating room conducted routine preoperative visits, they communicated effectively with the children and their families, and conducted psychological counseling. The visit time lasted nearly 30 minutes. On the day of surgery, all children were admitted to a special waiting room for children 0.5 h in advance, and venipuncture was performed by a circuit nurse. Colorful cartoon patterns were depicted on the walls of the waiting room, and various toys for children were placed indoors. After entering the operating room, the child was accompanied by a parent in the waiting room for the child to wait for surgery. During the period, a nurse in the research group gave routine psychological comfort, preoperative guidance, answered questions about anesthesia and surgery raised by the children and their parents. Before anesthesia induction, the child was brought into the operating room for anesthesia induction and surgery by operating room nurse, anesthesiologist, and surgeon, while the child's parents leave the waiting room and wait outside the operating room.

The researchers assessed the children's anxiety status, the degree of cooperation during the induction of anesthesia, and recorded the heart rate and blood pressure of the children at three moments: before entering the operating room (baselineT0), entering the operating room(T1), and before induction of anesthesia(T2).Before data collection, researchers who conducting data collection should be trained in measurement tools and assessment methods. The training contents mainly include: (1) explaining the purpose, meaning and the scoring method of the measurement tools; (2) Scoring the child's anxiety through pictures at three time points, discussing the reasons for consistent or inconsistent results, and repeating until the coefficient of agreement κ≥0.8.

ELIGIBILITY:
Inclusion Criteria:

* With age from 3 to 12 years old;
* Had normal mental, psychological and intellectual development;
* Must receive general anesthesia surgery;
* Must be volunteered to join the study.

Exclusion Criteria:

* Receive an emergency surgery;
* With unstable vital signs or critical illness.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 181 (Actual)
Dates: Start 2019-04-07 (Actual); Primary Completion 2019-06-08 (Actual); Study Completion 2019-10-06 (Actual)

PRIMARY OUTCOMES:
The change from T0(baseline) the scores of anxiety of change at T1( entering the operating room) | T0(before entering the operating room )--T1(entering the operating room)
  The outcome 1 was measured by Modified Yale Preoperative Anxiety Scale-Short Form（mYPAS -SF),it is an observational behavioral medical scale, which can be used in surgical children to assess the preoperative anxiety level. mYPAS included 5 parts (mental state, language, emotional expression, arousal state, and dependence on parents).Each item of the scale corresponds to a different score. During the evaluation, the children's behaviors correspond to the corresponding items. The children's behaviors are divided into 1-4 grades or 1-6 grades. After conversion, the total score is 22.92-100 point. The lower the score, the lower the anxiety level of the child, and vice versa.
The change from T1( entering the operating room)the scores of anxiety of change at T2(before induction of anesthesia) | T1(entering the operating room)--T2(before induction of anesthesia)
  The outcome 1 was measured by Modified Yale Preoperative Anxiety Scale-Short Form（mYPAS -SF),it is an observational behavioral medical scale, which can be used in surgical children to assess the preoperative anxiety level. mYPAS included 5 parts (mental state, language, emotional expression, arousal state, and dependence on parents).Each item of the scale corresponds to a different score. During the evaluation, the children's behaviors correspond to the corresponding items. The children's behaviors are divided into 1-4 grades or 1-6 grades. After conversion, the total score is 22.92-100 point. The lower the score, the lower the anxiety level of the child, and vice versa.
The degree of cooperation of children during anesthesia induction | T2(before induction of anesthesia)
  The outcome 2 was measured by the Induction Compliance Checklist , There are 11 items in total, with scores ranging from 0 to 10 points. A score of 0 points means that the induction was successful without any uncooperative behavior; 10 points mean that the induction failed, that is, the child was completely passive and the degree of cooperation was very poor. If the child has the same condition as the item on the scale, the child can get 1 point, and the points were added up to get the final total score. The lower the total score, the better the cooperation.
The change from T0(baseline) the heart rate of change at T1( entering the operating room) | T0(before entering the operating room )--T1(entering the operating room)
  The evaluation heart rate was performed by the same portable electronic sphygmomanometer (OMRON HEM-7124). The vital signs in the operation room were measured by the same ECG monitor (Minray BeneView T8).The heart rate was measured by beats per minute.
The change from T1( entering the operating room)the heart rate of change at T2(before induction of anesthesia) | T1(entering the operating room)--T2(before induction of anesthesia)
  The evaluation heart rate was performed by the same portable electronic sphygmomanometer (OMRON HEM-7124). The vital signs in the operation room were measured by the same ECG monitor (Minray BeneView T8).The heart rate was measured by beats per minute.
The change from T0(baseline) the systolic blood pressure of change at T1( entering the operating room) | T0(before entering the operating room )--T1(entering the operating room)
  The evaluation systolic blood pressure was performed by the same portable electronic sphygmomanometer (OMRON HEM-7124). The vital signs in the operation room were measured by the same ECG monitor (Minray BeneView T8). The systolic blood pressure was measured by mmHg.
The change from T1( entering the operating room)the systolic blood pressure of change at T2(before induction of anesthesia) | T1(entering the operating room)--T2(before induction of anesthesia)
  The evaluation systolic blood pressure was performed by the same portable electronic sphygmomanometer (OMRON HEM-7124). The vital signs in the operation room were measured by the same ECG monitor (Minray BeneView T8).The systolic blood pressure was measured by mmHg.
The change from T0(baseline) the diastolic blood pressure of change at T1( entering the operating room) | T0(before entering the operating room )--T1(entering the operating room)
  The evaluation diastolic blood pressure was performed by the same portable electronic sphygmomanometer (OMRON HEM-7124). The vital signs in the operation room were measured by the same ECG monitor (Minray BeneView T8).The diastolic blood pressure was measured by mmHg.
The change from T1( entering the operating room)the diastolic blood pressure of change at T2(before induction of anesthesia) | T1(entering the operating room)--T2(before induction of anesthesia)
  The evaluation diastolic blood pressure was performed by the same portable electronic sphygmomanometer (OMRON HEM-7124). The vital signs in the operation room were measured by the same ECG monitor (Minray BeneView T8).The diastolic blood pressure was measured by mmHg.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No
The process of data collection cost a lot of human and material resources, some of the data was privacy information of participants, and so on. Considering this, it is improper to share these data.

REFERENCES:
- [Background] Schneemilch CE, Bachmann H, Ulrich A, Elwert R, Halloul Z, Hachenberg T. Clonidine decreases stress response in patients undergoing carotid endarterectomy under regional anesthesia: a prospective, randomized, double-blinded, placebo-controlled study. Anesth Analg. 2006 Aug;103(2):297-302, table of contents. doi: 10.1213/01.ane.0000223673.68072.42. PMID 16861405
- [Background] Santiago AE, Issy AM, Sakata RK. Effects of preoperative intravenous clonidine in patients undergoing cataract surgery: a double-blind, randomized trial. J Ophthalmol. 2014;2014:346549. doi: 10.1155/2014/346549. Epub 2014 Sep 2. PMID 25276415
- [Background] Brans K, Koval P, Verduyn P, Lim YL, Kuppens P. The regulation of negative and positive affect in daily life. Emotion. 2013 Oct;13(5):926-39. doi: 10.1037/a0032400. Epub 2013 Jun 3. PMID 23731436
- [Background] Jallo N, Ruiz RJ, Elswick RK Jr, French E. Guided imagery for stress and symptom management in pregnant african american women. Evid Based Complement Alternat Med. 2014;2014:840923. doi: 10.1155/2014/840923. Epub 2014 Feb 25. PMID 24719646
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 Statement: updated guidelines for reporting parallel group randomised trials. BMC Med. 2010 Mar 24;8:18. doi: 10.1186/1741-7015-8-18. PMID 20334633
- [Background] Kain ZN, Mayes LC, Cicchetti DV, Bagnall AL, Finley JD, Hofstadter MB. The Yale Preoperative Anxiety Scale: how does it compare with a "gold standard"? Anesth Analg. 1997 Oct;85(4):783-8. doi: 10.1097/00000539-199710000-00012. PMID 9322455
- [Background] Jenkins BN, Fortier MA, Kaplan SH, Mayes LC, Kain ZN. Development of a short version of the modified Yale Preoperative Anxiety Scale. Anesth Analg. 2014 Sep;119(3):643-650. doi: 10.1213/ANE.0000000000000350. PMID 25010821
- [Result] Kain ZN, Caldwell-Andrews AA, Maranets I, McClain B, Gaal D, Mayes LC, Feng R, Zhang H. Preoperative anxiety and emergence delirium and postoperative maladaptive behaviors. Anesth Analg. 2004 Dec;99(6):1648-1654. doi: 10.1213/01.ANE.0000136471.36680.97. PMID 15562048
- [Result] Eijlers R, Dierckx B, Staals LM, Berghmans JM, van der Schroeff MP, Strabbing EM, Wijnen RMH, Hillegers MHJ, Legerstee JS, Utens EMWJ. Virtual reality exposure before elective day care surgery to reduce anxiety and pain in children: A randomised controlled trial. Eur J Anaesthesiol. 2019 Oct;36(10):728-737. doi: 10.1097/EJA.0000000000001059. PMID 31356373
- [Result] Meletti DP, Meletti JFA, Camargo RPS, Silva LM, Modolo NSP. Psychological preparation reduces preoperative anxiety in children. Randomized and double-blind trial. J Pediatr (Rio J). 2019 Sep-Oct;95(5):545-551. doi: 10.1016/j.jped.2018.05.009. Epub 2018 Jun 30. PMID 31340899
- [Result] Kumar A, Das S, Chauhan S, Kiran U, Satapathy S. Perioperative Anxiety and Stress in Children Undergoing Congenital Cardiac Surgery and Their Parents: Effect of Brief Intervention-A Randomized Control Trial. J Cardiothorac Vasc Anesth. 2019 May;33(5):1244-1250. doi: 10.1053/j.jvca.2018.08.187. Epub 2018 Aug 22. PMID 30243867
- [Result] Vagnoli L, Bettini A, Amore E, De Masi S, Messeri A. Relaxation-guided imagery reduces perioperative anxiety and pain in children: a randomized study. Eur J Pediatr. 2019 Jun;178(6):913-921. doi: 10.1007/s00431-019-03376-x. Epub 2019 Apr 3. PMID 30944985
- [Result] Aytekin A, Doru O, Kucukoglu S. The Effects of Distraction on Preoperative Anxiety Level in Children. J Perianesth Nurs. 2016 Feb;31(1):56-62. doi: 10.1016/j.jopan.2014.11.016. Epub 2015 Nov 11. PMID 26847781
- [Result] Millett CR, Gooding LF. Comparing Active and Passive Distraction-Based Music Therapy Interventions on Preoperative Anxiety in Pediatric Patients and Their Caregivers. J Music Ther. 2018 Jan 13;54(4):460-478. doi: 10.1093/jmt/thx014. PMID 29253180
- [Result] Atak M, Ozyazicioglu N. The Effect of Different Audio Distraction Methods on Children's Postoperative Pain and Anxiety. J Perianesth Nurs. 2021 Feb;36(1):75-80. doi: 10.1016/j.jopan.2020.06.028. Epub 2020 Oct 24. PMID 33531174
- [Result] Kuhlmann AYR, van Rosmalen J, Staals LM, Keyzer-Dekker CMG, Dogger J, de Leeuw TG, van der Toorn F, Jeekel J, Wijnen RMH, van Dijk M. Music Interventions in Pediatric Surgery (The Music Under Surgery In Children Study): A Randomized Clinical Trial. Anesth Analg. 2020 Apr;130(4):991-1001. doi: 10.1213/ANE.0000000000003983. PMID 30633058
- [Result] Chow CH, Van Lieshout RJ, Schmidt LA, Dobson KG, Buckley N. Systematic Review: Audiovisual Interventions for Reducing Preoperative Anxiety in Children Undergoing Elective Surgery. J Pediatr Psychol. 2016 Mar;41(2):182-203. doi: 10.1093/jpepsy/jsv094. Epub 2015 Oct 17. PMID 26476281
- [Result] Beizaee Y, Rejeh N, Heravi-Karimooi M, Tadrisi SD, Griffiths P, Vaismoradi M. The effect of guided imagery on anxiety, depression and vital signs in patients on hemodialysis. Complement Ther Clin Pract. 2018 Nov;33:184-190. doi: 10.1016/j.ctcp.2018.10.008. Epub 2018 Oct 17. PMID 30396619
- [Result] Kain ZN, MacLaren J, McClain BC, Saadat H, Wang SM, Mayes LC, Anderson GM. Effects of age and emotionality on the effectiveness of midazolam administered preoperatively to children. Anesthesiology. 2007 Oct;107(4):545-52. doi: 10.1097/01.anes.0000281895.81168.c3. PMID 17893449
- [Result] Bradt J, Dileo C, Shim M. Music interventions for preoperative anxiety. Cochrane Database Syst Rev. 2013 Jun 6;2013(6):CD006908. doi: 10.1002/14651858.CD006908.pub2. PMID 23740695
- [Derived] Wang X, Zhang J, Xin H, Tan W, Liu Y, Wan J. Effectiveness of two distraction strategies in reducing preoperative anxiety in children in China: A randomized controlled trial. J Pediatr Nurs. 2023 Jan-Feb;68:e8-e15. doi: 10.1016/j.pedn.2022.10.013. Epub 2022 Nov 17. PMID 36402600